CLINICAL TRIAL: NCT03430102
Title: Validation of the Indicor Device in Identifying Elevated Left Ventricular End Diastolic Pressure LVEDP
Brief Title: Indicor Validation
Status: Completed | Type: Observational
Sponsor: Vixiar Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00022390
Record Dates: First submitted 2018-01-29; First posted 2018-02-12 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- LeftHeartCath: Patients scheduled for LV catheterization for direct measurement of LVEDP
  Interventions: Diagnostic Test: Indicor

INTERVENTIONS:
Diagnostic Test: Indicor — Calculation of LVEDP via analysis of PPG waveform with Valsalva

SUMMARY:
The study is designed to repeat an initial training set study conducted at Johns Hopkins Medical Center, comparing a new investigational device, Indicor, a non-invasive tool for estimating left ventricular end diastolic pressure (LVEDP), to the gold standard, invasively measured LVEDP via direct measurement via left heart catheterization. The study is divided into an initial training set, followed by the validation set which is designed to support an FDA 510(k) submission and validate the final algorithm. Patients will be enrolled who are scheduled to undergo a cardiac catheterization and will be asked to perform three tests with the Indicor.

DETAILED DESCRIPTION:
Patients who are scheduled to undergo a left heart cardiac catheterization for direct measure of left ventricular end diastolic pressure (LVEDP) as part of routine care will be asked to participate. Investigators will take non-invasive measures of LVEDP using the Indicor device, repeated at three time points before and after the catheterization procedure. The Indicor indirectly measures LVEDP by calculating a value from finger photoplethysmography (PPG) waveforms that will be recorded while the patient performs a Valsalva maneuver.

Participants baseline characteristics will be gathered from the electronic medical record, including history of coronary artery disease, heart failure, hypertension, diabetes, or lung disease; list of blood pressure medications; serum markers of kidney function; and echocardiogram measurements including ejection fraction. These parameters will be used to assess relevance to the calculation of LVEDP by Indicor.

The first Indicor measure will be conducted before the catheterization procedure. PPG probes will be attached to participants' first or second finger. Participants will be asked to strain as if having a bowel movement (Valsalva maneuver) for 10 seconds. Participants will blow into a pressure transducer that measures and displays the pressure of their effort. The Indicor device will acquire 3 successful efforts.

During the cardiac catheterization, while the pressure transducer used by the clinical team to measure LVEDP is in the aorta, the Valsalva testing will be repeated. The device will again acquire 3 successful efforts. This will allow investigators to determine how well the amplitude changes of the PPG signal during Valsalva maneuver reflect the amplitude changes of central arterial pressure during the Valsalva maneuver. According to experienced catheterization cardiologists, this set of tests will not add significant risk to the procedure. This second set of tests may not be performed in all participants.

Immediately after the cardiac catheterization, while the patient is still on the catheterization table, the Valsalva testing will be repeated. The device will again acquire 3 successful efforts.

ELIGIBILITY:
Inclusion Criteria:

-Adult patients scheduled to undergo a left-heart catheterization that will include the measurement of left ventricular end-diastolic pressure (LVEDP)

Exclusion Criteria:

* Weight <88 pounds (40 kilograms)
* Atrial flutter or atrial fibrillation with an irregular ventricular response
* Significant atrial or ventricular ectopy
* History of paradoxical emboli
* Hypertrophic obstructive cardiomyopathy
* History of paradoxical emboli
* Known intracardiac shunt
* Known severe aortic valve stenosis or known severe mitral valve stenosis
* History of embolic cerebrovascular accident
* Clinically unstable
* Uncontrolled hypertension (systolic BP >160 mmHg or diastolic BP> 100 mmHg)
* Hypotension (systolic BP <90 mmHg)
* Symptomatic bradycardia
* Known cholesterol emboli
* Poor LV function with known LV thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo cardiac catheterization as part of their routine care and clinically indicated
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
C-LVEDP | During patients scheduled left heart cardiac catheterization
  Specificity of Calculated LVEDP (C-LVEDP) in identifying invasively Measured LVEDP (M-LVEDP) > 20 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Harry Silber, MD, PhD, Principal Investigator — Johns Hopkins Medical Center
Locations (4):
- United States (4):
  - Christiana Care, Newark, Delaware
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Stony Brook Medicine, Stony Brook, New York
  - Lancaster General Health, Lancaster, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilotra NA, Tedford RJ, Wittstein IS, Yenokyan G, Sharma K, Russell SD, Silber HA. Usefulness of Pulse Amplitude Changes During the Valsalva Maneuver Measured Using Finger Photoplethysmography to Identify Elevated Pulmonary Capillary Wedge Pressure in Patients With Heart Failure. Am J Cardiol. 2017 Sep 15;120(6):966-972. doi: 10.1016/j.amjcard.2017.06.029. Epub 2017 Jun 28. PMID 28754567
- [Background] Galiatsatos P, Win TT, Monti J, Johnston PV, Herzog W, Trost JC, Hwang CW, Fridman GY, Wang NY, Silber HA. Usefulness of a Noninvasive Device to Identify Elevated Left Ventricular Filling Pressure Using Finger Photoplethysmography During a Valsalva Maneuver. Am J Cardiol. 2017 Apr 1;119(7):1053-1060. doi: 10.1016/j.amjcard.2016.11.063. Epub 2017 Jan 5. PMID 28185634
- [Background] Silber HA, Trost JC, Johnston PV, Maughan WL, Wang NY, Kasper EK, Aversano TR, Bush DE. Finger photoplethysmography during the Valsalva maneuver reflects left ventricular filling pressure. Am J Physiol Heart Circ Physiol. 2012 May 15;302(10):H2043-7. doi: 10.1152/ajpheart.00609.2011. Epub 2012 Mar 2. PMID 22389389
- [Background] Sharma GV, Woods PA, Lambrew CT, Berg CM, Pietro DA, Rocco TP, Welt FW, Sacchetti P, McIntyre KM. Evaluation of a noninvasive system for determining left ventricular filling pressure. Arch Intern Med. 2002 Oct 14;162(18):2084-8. doi: 10.1001/archinte.162.18.2084. PMID 12374516
- [Background] Gillard C, Henuzet C, Lallemand J, Moscariello A, Guillaume M, Van Meerhaeghe A. Operating characteristics of the Finapress system to predict elevated left ventricular filling pressure. Clin Cardiol. 2006 Mar;29(3):107-11. doi: 10.1002/clc.4960290305. PMID 16596832
- [Background] Zema MJ. Bedside assessment of cardiac hemodynamics: role of the simple Valsalva maneuver. Am J Med. 2012 Aug;125(8):e13; author reply e15-6. doi: 10.1016/j.amjmed.2011.12.020. No abstract available. PMID 22840672
- [Background] Felker GM, Cuculich PS, Gheorghiade M. The Valsalva maneuver: a bedside "biomarker" for heart failure. Am J Med. 2006 Feb;119(2):117-22. doi: 10.1016/j.amjmed.2005.06.059. PMID 16443410
- [Background] Stevenson LW, Perloff JK. The limited reliability of physical signs for estimating hemodynamics in chronic heart failure. JAMA. 1989 Feb 10;261(6):884-8. PMID 2913385